CLINICAL TRIAL: NCT02439814
Title: Effect of Pregnenolone on Cue-reactivity in Marijuana-dependent Individuals
Brief Title: Pregnenolone and Marijuana Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO42135
Record Dates: First submitted 2015-04-22; First posted 2015-05-12 (Estimated); Results first posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Marijuana Dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregnenolone (Experimental)
  Interventions: Drug: Pregnenolone
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pregnenolone — Pregnenolone is a steroid that occurs naturally in the body, and early studies have shown that pregnenolone may block the effects of marijuana intoxication
  Arms: Pregnenolone
Other: Placebo — Inactive comparator
  Arms: Placebo

SUMMARY:
The cannabinoid delta 9-tetrahydrocannabinol (THC) is the primary psychoactive component of marijuana. THC is believed to be a significant factor in the addictive potential associated with marijuana use. In addition, attenuated levels of endogenous endocannabinoids have been found in alcohol-dependent individuals as compared to social drinkers, suggesting that changes in the sensitivity of the endogenous endocannabinoid system play a role in the transition from recreational drug use to substance use disorders. Thus, pharmacotherapies that target the cannabinoid system may be effective strategies for reducing marijuana use and dependence. Recent preclinical data demonstrate that the neurosteroid pregnenolone (PREG) inhibits THC activation of cannabinoid receptors and decreases symptoms of marijuana intoxication. In addition, other studies show that PREG inhibits drug-seeking behavior. This pilot study will provide important preliminary data on the effect of an acute dose of PREG on cue-related craving in individuals with cannabis use disorder.

DETAILED DESCRIPTION:
Overview Thirty participants between the ages of 18 and 65 who meet DSM-V criteria for current for cannabis use disorder will complete a study visit. Participants will be randomized to receive either PREG (400 mg) (n=15) or placebo (PBO) (n=15). Two-hours after medication administration, the participants will complete a cue reactivity session. Blood samples will be collected prior to medication, post-medication and after the cue-reactivity session. The blood samples will be assayed for endogenous PREG and endocannabinoid levels. Subjective craving and mood data will also be collected.

Subjects Participants will be 30 men or women between the ages of 18 and 65 years who meet DSM-V criteria for cannabis use disorder. Additional inclusion criteria include use of acceptable methods of birth control if female and of childbearing potential, positive urine drug screen for cannabinoids at screening, consent to random assignment, and ability to read and provide informed consent. Exclusion criteria include women who are pregnant, nursing, or plan to become pregnant during the course of the study; having a history of or current psychotic disorder, bipolar disorder, or eating disorder; posing a current suicidal or homicidal risk; having evidence or history of serious medical disease; requiring concomitant therapy with psychotropic medication; being currently dependent on other substances, with the exception of nicotine; and patients who, in the investigator's opinion, would be unable to comply with study procedures or assessments.

Procedures

1. Recruitment. Subjects will be primarily recruited through media advertisements. The investigators have an active recruitment network in place, and have been able to consistently surpass recruitment goals even with concomitantly recruiting studies in this population, averaging enrollment of 11 participants per month. As such, the investigators do not anticipate any issues with successfully recruiting for this study in the proposed timeframe.
2. Screening/Assessment. Individuals will be initially screened for eligibility over the telephone by a trained research assistant. Major inclusion/exclusion criteria will be assessed during the phone interview, and if an individual seems potentially eligible, (s)he will be invited for an in-person interview with a member of the research team. Prior to any study procedures being performed, the individual will sign an IRB-approved informed consent form. A battery of standardized assessments will then be delivered (described below). A general medical history and physical exam will also be performed to ensure that the subject is eligible to participate. In the event that a patient is found to be ineligible to participate in this research protocol, he or she will be given an appropriate referral for further medical care or to an appropriate treatment program.
3. Session Preparation. The test session will be conducted at the MUSC Research NEXUS. Prior to leaving the assessment visit, participants will be instructed to avoid caffeine and marijuana on the day of the study visit. Participants will also be instructed to abstain from other drug (including alcohol) use for the three days prior to the study visit.
4. Study Visit. Participants will present to the Addiction Sciences Division at 12:00 on the day of the study visit. Female participants will complete a urine pregnancy test. If the results are negative, or if the participant is male, the subject will be breathalyzed and will provide a urine sample, which will be tested for the presence of cocaine, opiates, benzodiazepines, THC, and stimulants. If either test is positive for alcohol or any drug with the exception of marijuana, the study visit will be rescheduled. A saliva sample to test for drugs of abuse will also be collected. Nicotine patches will be provided to cigarette smokers to avoid nicotine withdrawal. Participants will be escorted to the MUSC Research NEXUS by study personnel. At 12:30, a blood sample will be collected from each participant. Each participant will also be asked to rate their craving and mood (described below). Medication will be administered to the participants by NEXUS personnel. Each participant will remain in a private room for two hours. At 2:30 a second blood sample will be collected from each participant and subjective ratings will be obtained. After the blood draw, study personnel will provide the participant with standardized cue-exposure instructions, stating that two sets of items will be presented and audio will be played through headphones. Control cues will be presented to each participant. Examples of these cues include a note pad, pencil, marker, cotton swabs and teabags.Wood chips will be presented as an olfactory cue and an auditory script will be played in which each participant will be asked to imagine a day at the beach. A third blood sample will be drawn and the participant will be asked to rate their craving and mood. Afterwards each participant will be presented with the marijuana cues. Examples of these cues include, blunt wrap, rolling papers, pipes, a pipe cleaner, small bag containing fake marijuana, an ashtray, a water bong and a fake joint. A marijuana stick cigarette and/or marijuana scented oil will be burned presented as an olfactory cue and each participant will listen to a script prompting recall of a recent pleasant experience with marijuana. Dr. McRae-Clark has a Schedule I DEA license, and has obtained marijuana for clinical trial use from NIDA. The investigators' laboratory and others have used these procedures to evoke craving in marijuana-dependent individuals [11, 12]. Blood samples and subjective ratings will be collected immediately, 15 minutes, 30 minutes and 60 minutes after the start of the marijuana cue session. After the final assessment each participant will be debriefed and compensated. In the event that a participant's craving remains elevated, he or she will be asked to remain in the NEXUS until their craving has subsided.

ELIGIBILITY:
General Inclusion / Exclusion Criteria Inclusion Criteria

1. Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Subjects must meet DSM-5 criteria for current cannabis use disorder (within the past three months). While individuals may endorse use of other substances, they must identify marijuana as their primary substance of abuse and must not meet criteria for any other substance use disorder (except nicotine) within the last 60 days. Due to the high comorbidity of marijuana and alcohol use disorder, subjects who meet criteria for mild alcohol use disorder will be included.
3. Subjects must consent to remain abstinent from alcohol for 24 hours and other drugs of abuse (except nicotine and marijuana) for three days immediately prior to the study visit. Subjects must abstain from marijuana for 24 hours prior to the study visit. By restricting marijuana use as proposed, subjects should not be under the acute effects of marijuana.
4. Subjects must consent to random assignment.

Exclusion Criteria

1. Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
2. Individuals taking exogenous gonadal steroids including estrogens, progestins and testosterone. This includes hormonal contraception and replacement therapy.
3. Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, neurological disease including diabetes or cancer, as these conditions may affect study outcomes.
4. Subjects with a history of or current psychotic disorder or bipolar affective disorder as these may interfere with subjective measurements.
5. Subjects taking any psychotropic medications, including SRI's or other antidepressants, opiates or opiate antagonists because these may affect test response. Individuals who take stimulants for treatment of ADHD will be allowed to participate.
6. Subjects with any acute illness or fever. Individuals who otherwise meet study criteria will be rescheduled for evaluation for participation.
7. Subjects who are unwilling or unable to maintain abstinence from alcohol and marijuana for 24 hours and other drugs of abuse (except nicotine) for three days prior to the study visit.
8. Subjects meeting DSM-5 criteria for a substance use disorder (other than nicotine, marijuana, or alcohol) within the past 60 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee McRae-Clark, PharmD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were primarily recruited through media advertisements and word of mouth.
Period: Overall Study
Arm/Group | Pregnenolone | Placebo
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnenolone | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 26.4 [19 to 49] | 25.6 [19 to 36] | 26 [19 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Subjective Rating of Marijuana Craving on 1-7 Likert Scale
Description: Change in craving from post medication administration to post active cue. Scale of 1-7 with 7 meaning the craving is most severe.
Time Frame: 12:40 to 14:45 (post med administration, post Marijuana cue
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 11 | 10
units on a scale | 1.64 (1.71) | 0.80 (1.79)

ADVERSE EVENTS:
Arm/Group | Pregnenolone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes